CLINICAL TRIAL: NCT00377325
Title: Cyclosporine in the Pharmacotherapy of Psoriasis
Brief Title: The Effectiveness of Lower Cyclosporine Doses for Psoriasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by the DSMB due to low recruitment
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Francisco Tausk, Professor, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AR050100 (NIH); R01AR050100 (NIH); NIH-7R01AR050100
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive full dose cyclosporin.
  Interventions: Drug: Cyclosporine
- 2 (Experimental): Participants will receive active drug full dose until cleared, then one dose every 4 days.
  Interventions: Drug: Cyclosporine
- 3 (Placebo Comparator): Participants will receive active drug full dose until clear, then full dose every 4 days with placebo on the intervening days.
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Cyclosporine — 4 mg/Kg/day; daily; liquid form; 6 months

SUMMARY:
This study will evaluate whether lower doses of cyclosporine can cause fewer side effects and still produce the same beneficial results that are seen with a standard cyclosporine dose regimen when treating individuals with moderate to severe psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory skin disease. It is believed to be caused by an overactive immune system that speeds the growth of skin cells. This abnormal skin growth results in patches of inflamed skin, which can itch, crack, and bleed. Cyclosporine is an immunosuppressant drug that is used in more severe cases of psoriasis to slow down the growth of skin cells. However, cyclosporine use is associated with several side effects, including kidney damage, high blood pressure, and skin sensitivity. This study will evaluate whether lower doses of cyclosporine can cause fewer side effects and still produce the same beneficial results that are seen with the standard administration of cyclosporine.

Participants in this study will receive treatment with cyclosporine for up to 30 weeks. Study visits will occur every 2 weeks and will include a physical exam, a psoriasis symptom evaluation, blood collection, and various questionnaires on quality-of-life issues. Participants will be followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Good health
* Exception that has been resistant to psoralen and ultraviolet A radiation (PUVA), methotrexate, and retinoids
* Moderate to severe, stable plaque psoriasis
* Normal organ and marrow function
* HIV uninfected

Exclusion Criteria:

* Topical therapy within 4 weeks of study entry
* Use of systemic, intralesional, or phototherapy within 1 year of study entry
* Use of cyclosporine in the past or use of other immunosuppressive medication within 6 months of study entry
* Inability to be followed or monitored regularly on a weekly basis
* Poorly controlled hypertension
* Severe infection, internal malignancy, immunodeficiency, gout, or liver disease
* Received more than 1,000 treatments of ultraviolet A (UVA)
* History of allergic reaction attributed to compounds of similar chemical or biological composition to cyclosporine
* Uncontrolled active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia that would limit study participation
* Women of childbearing potential and men unwilling to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of the study
* Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Improvement in psoriasis symptoms | Measured every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Tausk, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Department of Dermatology, Rochester, New York, United States